CLINICAL TRIAL: NCT00125385
Title: Phase I, Open-Label, Multi-Center, Single-Dose, Dose-Escalating, Safety, Tolerability and Pharmacokinetic of GC1008 in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Study of GC1008 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC100800103
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF; Idiopathic; Pulmonary; Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Fibrosis | interventions — fresolimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): Dose group
  Interventions: Biological: GC1008
- Cohort 2 (Experimental): Dose Group
  Interventions: Biological: GC1008
- Cohort 3 (Experimental): Dose Group
  Interventions: Biological: GC1008
- Cohort 4 (Experimental): Dose Group
  Interventions: Biological: GC1008
- Cohort 5 (Experimental): Dose Group
  Interventions: Biological: GC1008

INTERVENTIONS:
Biological: GC1008 — 0.3 mg/kg, IV on Day 0 and return to the clinic on 3,7, 10, 14, 21, 28, 42, 56, 84, 112, 140 post infusion for safety follow-up.
  Arms: Cohort 1
Biological: GC1008 — 1.0 mg/kg, IV on Day 0 and return to the clinic on 3,7, 10, 14, 21, 28, 42, 56, 84, 112, 140 post infusion for safety follow-up.
  Arms: Cohort 2
Biological: GC1008 — 2.0 mg/kg, IV on Day 0 and return to the clinic on 3,7, 10, 14, 21, 28, 42, 56, 84, 112, 140 post infusion for safety follow-up.
  Arms: Cohort 3
Biological: GC1008 — 4.0 mg/kg, IV on Day 0 and return to the clinic on 3,7, 10, 14, 21, 28, 42, 56, 84, 112, 140 post infusion for safety follow-up.
  Arms: Cohort 4
Biological: GC1008 — 8.0 mg/kg, IV on Day 0 and return to the clinic on 3,7, 10, 14, 21, 28, 42, 56, 84, 112, 140 post infusion for safety follow-up.
  Arms: Cohort 5

SUMMARY:
This study is designed to investigate whether GC1008, an antibody that neutralizes TGFb, is safe in treating patients with idiopathic pulmonary fibrosis. The highest dose without excessive side effects will be identified. Tests will determine how long GC1008 is in the body and how it is excreted.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent prior to any study-related procedures.
* Patients should have an established diagnosis of IPF.
* Pulmonary Function Tests (PFTs): FVC ≥ 50% and DLCO ≥ 25% of normal predicted values.
* Able to walk at least 500 feet (150 meters) during the 6-minute Walk Test (6MWT). During the 6MWT the patient must not require greater than 51/min supplemental oxygen to maintain oxygen saturation > 80%

Exclusion Criteria:

* Women who are pregnant or lactating; or who plan to become pregnant within 9 months after the infusion.
* Women of childbearing potential or men who are considering fathering a child unless taking medically acceptable contraceptive precautions;
* History of clinically significant environmental exposure, including dust, molds, asbestos, pigeons or other birds that may result in interstitial lung disease, or ingestion of a drug known to cause pulmonary fibrosis such as bleomycin.
* History of clinically significant respiratory diseases other than IPF.
* History of clinically significant cardiac, hepatic, or renal disease.
* History of cancer, precancerous state (e.g. familial polyposis, BRCA1, BRCA2), other than non-melanomatous skin cancer, within 5 years prior to Screening.
* Use of any investigational drug administered as part of a clinical trial within 12 weeks before Screening.
* Other pathology that might interfere with the assessment of the safety or efficacy of the test article.
* Other clinically significant, uncontrolled medical condition that, in the Investigator's opinion, might interfere with the assessment or follow-up.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To evaluate safety, tolerability, and pharmacokinetics (PKs) of single intravenous (IV) infusions of GC1008 in patients with IPF | up to 3 years

SECONDARY OUTCOMES:
To evaluate potential clinical outcomes and bioactivity of GC1008 | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- United States (7):
  - Denver, Colorado
  - Chicago, Illinois
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Nashville, Tennessee
  - Seattle, Washington
- Belgium, Belgium

REFERENCES:
- [Derived] Shenderov K, Collins SL, Powell JD, Horton MR. Immune dysregulation as a driver of idiopathic pulmonary fibrosis. J Clin Invest. 2021 Jan 19;131(2):e143226. doi: 10.1172/JCI143226. PMID 33463535